CLINICAL TRIAL: NCT01670929
Title: Pr-conceptional Progesterone for Unexplained Recurrent Miscarriage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, M D, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPROURM
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Abortion, Habitual
Keywords: recurrent miscarriages; progesterone
MeSH Terms: conditions — Abortion, Habitual | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone group (Active Comparator): progesterone (400 mg pessary, once daily)
  Interventions: Drug: Progesterone
- Placebo group (Placebo Comparator): Placebo (pessary, once daily)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Progesterone
  Arms: Progesterone group
Other: Placebo
  Arms: Placebo group

SUMMARY:
In women with unexplained recurrent miscarriages, progesterone (400 mg pessaries, twice daily), started soon as possible at luteal phase and after a positive pregnancy test and continued to 28 weeks of gestation, compared to placebo, ).

DETAILED DESCRIPTION:
Progesterone improves secondary outcomes such as gestation at delivery, on-going pregnancy at 12 weeks, survival at 28 days of neonatal life.

. Progesterone, compared to placebo, does not incur substantial adverse effects to the mother or the neonate.

Explore differential or subgroup effects of progesterone in prognostic subgroups.

. Perform an economic evaluation for cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Women with unexplained recurrent miscarriages (2 or more consecutive first trimester miscarriages).
2. Age 18-39 years at randomisation (likelihood of miscarriages due to chromosomal aberrations is higher in older women; such miscarriages are unlikely to be prevented by progesterone therapy).
3. Spontaneous conception (as confirmed by urinary pregnancy tests).
4. Willing and able to give informed consent.

Exclusion Criteria:

1. Age less than twenty or above forty years old.
2. Antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies [IgG or IgM]); other recognised thrombophilic conditions (testing according to usual clinic practice)
3. Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
4. Fibroids distorting uterine cavity.
5. Abnormal parental karyotype.
6. Other identifiable causes of recurrent miscarriages (tests initiated only if clinically indicated) e.g., diabetes, thyroid disease and systemic lupus erythematosus (SLE).

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of patients continued the pregnancy beyond 20 weeks gestation. | 2 years

SECONDARY OUTCOMES:
Number of miscarriages | 2 years

OTHER OUTCOMES:
Number of Live Birth | 2 years
Number of preterm delivery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M D, Principal Investigator — Faculity of medicine,Assiut university
Locations (1):
- Women's Health Hospital, Asyut, Egypt